CLINICAL TRIAL: NCT04472039
Title: Intraretinal Cystoid Changes After Vitrectomy With Membrane Peeling
Status: Completed | Type: Observational
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prof. Dr. Oliver Findl, MBA, Vienna Institute for Research in Ocular Surgery
Other Study IDs: RAC
Record Dates: First submitted 2020-07-11; First posted 2020-07-15 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Macular Edema, Cystoid
MeSH Terms: conditions — Macular Edema | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Studygroup: Retrospective analysis of OCT, IOP and distance corrected visual acuity from the patients history.
  Interventions: Device: optical coherence tomography (OCT)

INTERVENTIONS:
Device: optical coherence tomography (OCT) — OCT visualizes the retinal layers by backreflection of light

SUMMARY:
Aim of the study is to assess the rate of postoperative intraretinal cystoid changes after pars plana vitrectomy with membrane peeling and peribulbar application of triamcinolone acetonide and to examine possible risk factors for postoperative intraretinal cystoid changes.

DETAILED DESCRIPTION:
Epiretinal membranes (ERM) are disorders leading to vision loss and metamorphopsia. Vitrectomy with membrane peeling has developed to be the gold-standard in treatment of ERM. Nevertheless, there are about 10% of patients having intraretinal cystoid changes after surgery with potential for disturbance of visual acuity. The aim of the study is to assess the rate of postoperative intraretinal cystoid changes after pars plana vitrectomy with membrane peeling and peribulbar application of triamcinolone acetonide and to examine possible risk factors for postoperative intraretinal cystoid changes.

ELIGIBILITY:
Inclusion Criteria:

* presence of an ERM
* indication for membrane peeling defined as significant loss of vision and/or metamorphopsia due to the ERM
* application of periocular triamcinolone acetonide at the end of surgery
* at least one follow-up examination present in the patient's history

Exclusion Criteria:

* macular edema caused by conditions other than ERM (such as choroidal neovascularization, diabetic macular edema, etc.)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients having undergone pars plana vitrectomy with membrane peeling and periocular application of triamcinolone acetonide at the end of surgery between June 2019 and January 2020 at the department of Ophthalmology of the Hanusch Hospital in Vienna, Austria, were selected for the study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Intraretinal cystoid changes | 3 months
  presence of intraretinal cystoid changes in OCT is assessed during the time period of 3 months after surgery

SECONDARY OUTCOMES:
intraocular pressure (IOP) | 3 months
  intraocular pressure is examined during the time period of 3 months after surgery
distance corrected visual acuity | 3 months
  distance corrected visual acuity is measured at baseline and 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prof., Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna, Vienna, Austria